CLINICAL TRIAL: NCT02752373
Title: A Health Economic Study Evaluating the Brain Sentinel® GTC Seizure Detection and Information Systems Impact on Epilepsy and Healthcare Utilization
Status: Terminated | Type: Observational
Why Stopped: This study was terminated due to low enrollment
Sponsor: Brain Sentinel (Other)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HE-1.5-03.2016
Record Dates: First submitted 2016-03-28; First posted 2016-04-27 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Epilepsy
Keywords: GTC Seizures
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Brain Sentinel Seizure Detection and Information System — The Brain Sentinel® GTC Seizure Detection and Information System is an ambulatory system designed to continuously monitor and perform real-time analysis of surface electromyography (sEMG) data to detect GTC seizures and to provide an alarm to alert caregivers within 30 seconds of bilateral, appendicular, tonic extension that a seizure is occurring. The System is for recording and storing sEMG data, which is subsequently reviewed by a trained healthcare professional in the outpatient clinical setting. The Brain Sentinel® GTC Seizure Detection and Information System is intended for real time monitoring of pediatric and adult patients who have an arm circumference ranging from at least 16 cm to no greater than 51 cm at the biceps. It may be used in the home or healthcare facilities for real-time monitoring during the day, night, or for continuous monitoring, including during the titration of, or the withdrawal from anti-epileptic drugs.

SUMMARY:
This is an open label prospective study of the impact on healthcare utilization of a surface Electromyography (sEMG) based seizure detection system for detecting Generalized Tonic-Clonic (GTC) Seizures.

DETAILED DESCRIPTION:
The Brain Sentinel® GTC Seizure Detection and Information System is an ambulatory system designed to continuously monitor and perform real-time analysis of surface electromyography (sEMG) data to detect GTC seizures and to provide an alarm to alert caregivers within 30 seconds of bilateral, appendicular, tonic extension that a seizure is occurring. The System is for recording and storing sEMG data, which is subsequently reviewed by a trained healthcare professional in the outpatient clinical setting. The Brain Sentinel® GTC Seizure Detection and Information System is intended for real time monitoring of pediatric and adult patients who have an arm circumference ranging from at least 16 cm to no greater than 51 cm at the biceps. It may be used in the home or healthcare facilities for real-time monitoring during the day, night, or for continuous monitoring, including during the titration of, or the withdrawal from anti-epileptic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a history of GTC seizures, either primary GTC or partial onset seizures with secondary generalization
* Male or female greater than 2 years of age
* Has an upper arm circumference which is adequate for proper fit of the EMG monitor (at least 16-51 cm)
* Be able to tolerate wearing the device on the upper arm
* Can understand and sign written informed consent, or will have a parent or a legally authorized representative (LAR) who can do so, prior to the performance of any study assessments
* Subject and/or Primary Caregiver must be competent to follow all study procedures.
* Is able to read, speak and understand English
* At least 2 or more Emergency Department visits in the previous 12 months for seizure related care

Exclusion Criteria:

* The subject is homeless or in a home without a power supply.
* The subject is allergic to adhesives or any component of the electrode patch assembly.
* The subject self-reports that she is pregnant or planning to become pregnant while using the device.

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with a history of GTC seizures, either primary GTC or partial onset seizures with secondary generalization
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2016-05; Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Evaluate the change in associated healthcare costs for patients with a GTC seizure detection and information system | 12 months prior to receiving the device and at 2 months and after 6 months of device use
  Evaluate the change in associated healthcare costs for patients 12 months prior as compared to 2 months and each 6 months of system use and compared to a similar population of epilepsy patients.

SECONDARY OUTCOMES:
Evaluate impact on healthcare utilization for patients with a GTC seizure detection and information system in the form of the change of the number of Emergency Department Visits | 12 months prior to receiving the device and at 2 months and after 6 months of device use
  The change in number of Emergency Department visits will be compared between the 12 months prior to receiving the device and at 2 months and after 6 months of device use.
Evaluate impact on healthcare utilization for patients with a GTC seizure detection and information system in the form of the change in number of inpatient hospitalizations | 12 months prior to receiving the device and at 2 months and after 6 months of device use
  The change in number of inpatient hospitalizations will be compared between the 12 months prior to receiving the device and at 2 months and after 6 months of device use.
Evaluate impact on healthcare utilization for patients with a GTC seizure detection and information system in the form of the change in number of EEGs | 12 months prior to receiving the device and at 2 months and after 6 months of device use
  The change in number of EEGs will be compared between the 12 months prior to receiving the device and at 2 months and after 6 months of device use.
Evaluate impact on healthcare utilization for patients with a GTC seizure detection and information system in the form of the change in number of Long Term Video EEG Monitoring (LTM) | 12 months prior to receiving the device and at 2 months and after 6 months of device use
  The change in number of Long Term Video EEG Monitoring (LTM) will be compared between the 12 months prior to receiving the device and at 2 months and after 6 months of device use.
Evaluate impact on healthcare utilization for patients with a GTC seizure detection and information system in the form of the change in number of outpatient clinic visits in patients | 12 months prior to receiving the device and at 2 months and after 6 months of device use
  The change in number of outpatient clinic visits in patients will be compared between the 12 months prior to receiving the device and at 2 months and after 6 months of device use.
Evaluate impact on healthcare utilization for patients with a GTC seizure detection and information system in the form of the change in number of no-shows and/or patient cancellations | 12 months prior to receiving the device and at 2 months and after 6 months of device use
  The change in number of no-shows and/or patient cancellations will be compared between the 12 months prior to receiving the device and at 2 months and after 6 months of device use.
Evaluate impact on healthcare utilization for patients with a GTC seizure detection and information system by assessing the change in seizure frequency for each type (reported as per month) | 12 months prior to receiving the device and at 2 months and after 6 months of device use
  Change in seizure frequency for each type (reported as per month) will be compared between the 12 months prior to receiving the device and at 2 months and after 6 months of device use.
Evaluate impact on healthcare utilization for patients with a GTC seizure detection and information system by assessing change in epilepsy etiology (including, but not limited to a new diagnosis of psychogenic non-epileptic spells) | 12 months prior to receiving the device and at 2 months and after 6 months of device use
  Change in epilepsy etiology (including, but not limited to a new diagnosis of psychogenic non-epileptic spells) will be compared between the 12 months prior to receiving the device and at 2 months and after 6 months of device use.
Evaluate impact on healthcare utilization for patients with a GTC seizure detection and information system by assessing clarification of diagnosis | 12 months prior to receiving the device and at 2 months and after 6 months of device use
  Clarification of diagnosis, if applicable, will be compared between the 12 months prior to receiving the device and at 2 months and after 6 months of device use.
Evaluate impact on healthcare utilization for patients with a GTC seizure detection and information system by assessing change in epilepsy treatment | 12 months prior to receiving the device and at 2 months and after 6 months of device use
  Change in epilepsy treatment will be compared between the 12 months prior to receiving the device and at 2 months and after 6 months of device use.
To evaluate the impact of epilepsy on families and patients ages > 11 receiving Brain Sentinel® System | 12 months prior to receiving the device and at 2 months and after 6 months of device use
  Assess data captured on Impact on Families questionnaire collected at baseline, 2 months, and each 6 month time period during use of the device.
To evaluate the change in quality of life for patients ages > 11 receiving Brain Sentinel® System | 12 months prior to receiving the device and at 2 months and after 6 months of device use
  Assess data captured on Quality of Life in Epilepsy questionnaire collected at baseline, 2 months, and each 6 month time period during use of the device.

CONTACTS AND LOCATIONS:
Overall Officials: Anup Patel, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No